CLINICAL TRIAL: NCT05738551
Title: Obez Bireylerde Kan Alma esnasında Uygulanan Iki farklı Nonfarmakolojik yöntemin ağrı ve kaygı üzerine Etkisinin Incelenmesi Randomize kontrollü çalışma
Brief Title: Non-pharmacolytic Method in Obese; Pain and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Rukiye Burucu, Assit. Prof., Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HİLAL
Record Dates: First submitted 2023-01-23; First posted 2023-02-22 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Obesity
Keywords: obesity; pain; anxiety; vascular access
MeSH Terms: conditions — Obesity; Pain; Anxiety Disorders | interventions — Chewing Gum

STUDY DESIGN:
Intervention Model Description: Three-arm randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STRESS BALL (Experimental): Starting 5 minutes before the access to the vascular access, the patient will be asked to squeeze the stress ball in the palm until the blood collection is completed.
  Interventions: Other: stress ball
- CHEWİNG GUM (Experimental): Starting 5 minutes before the vascular access, the patient will be allowed to chew gum until the blood collection is completed.
  Interventions: Other: chewing gum
- ROUTINE APPLICATION (No Intervention): Only within the scope of routine practice of the patient, vascular access will be provided and the blood collection process will be completed.

INTERVENTIONS:
Other: stress ball — Applicable to group 1
  Arms: STRESS BALL
Other: chewing gum — Applicable to group 2
  Arms: CHEWİNG GUM

SUMMARY:
Access to the vascular access is difficult in obese patients. Therefore, vascular access can be challenging and worrying for obese individuals. This strain causes pain and anxiety. Different interventions can be applied to reduce the pain and anxiety felt. One of them is the methods of distraction. Among these methods, chewing gum and using a stress ball can contribute positively to the pain and anxiety at the entrance to the vein in order to draw blood in obese individuals. In addition, these interventions may affect vital parameters. It was aimed to evaluate the effects of chewing gum and using a stress ball during vascular access in obese individuals on pain level, anxiety level and vital signs

DETAILED DESCRIPTION:
It is a three-armed randomized controlled trial.

Research Questions/Hypotheses:

H1: There is a difference between the arterial blood pressure, heart rate and oxygen saturation values of the groups H2: There is a difference between the state anxiety scores of the groups H3: There is a difference between the pain scores experienced by the groups

Type of Research:

3 groups post-test Randomized controlled trial

Location and Features of the Research:

The research will be completed in the outpatient blood collection unit of XXX hospital.

The populaıon of the Research:

The population of the research will be the patients who applied to the blood collection unit of XXX hospital.

Sample of the Research:

The sample of the research; An effect size of 0.35 was calculated as 108 with a margin of error 0.05 and a power of 0.90.

F tests - ANOVA: Fixed effects, omnibus, one-way Analysis: A priori: Compute required sample size Input: Effect size f = 0.35 α err prob = 0.05 Power (1-β err prob) = 0.90 Number of groups = 3 Output: Noncentrality parameter λ = 13.2300000 Critical F = 3.0828520 Numerator df = 2 Denominator df = 105 Total sample size = 108 Actual power = 0.9047332

Randomization A random.org package program was used for randomization, and a randomization table was created (Random.Org).

In the study, the patient, the nurse who took blood and the researcher will not be blinded, the people who made the randomization and statistics and the person who collected the data after the intervention will be blinded.

Inclusion Criteria for Participants in the Study:

* Being over 18 years old
* Having a body mass index of 30 and above
* Giving blood for analyzes upon the request of the physician
* Having the harmony of place and time
* Willingness to participate in the research Exclusion criteria
* Absence of vision and hearing problems
* Presence of any disease that may affect pain perception
* Having cognitive problems
* Having a condition that prevents chewing gum
* Having a condition that prevents him from using the stress ball

Data Collection Tools:

Individual identification form, Visual comparison scale (VAS), state anxiety inventory, pulse oximeter, sphygmomanometer, tape measure Individual introduction form and initiative materials It is a form consisting of 12 questions prepared by researchers in accordance with the literature. It includes the socio-demographic and health-related characteristics of individuals.

VAS (Visual Comparison Scale) The scale consists of or vertical lines. The scale is scaled to 10 cm/100 mm. Horizontal form will be used in this study. A score of 0 on the scale in the assessment of pain indicates that there is no pain during the blood draw procedure, and a score of 10 indicates unbearable/very severe pain.

State Anxiety Inventory It was developed by Spielberg et al (1964). Öner and le Compte (1983) was adapted into Turkish. It can measure state and trait anxiety separately, a total of 40 items. In this study, only the 20-item section that measures state anxiety will be used. It gives information about the individual's feelings only at that moment. It is a four-point Likert-type scale; It is evaluated as "not at all", "somewhat", "a lot" and "completely" with 1, 2, 3 and 4 points. In the state anxiety scale, items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reversed items. The scale scores between 20 and 80, with a high score indicating a high level of anxiety. However, since the scale is not calculated straight, it is stated that the average score generally varies between 36-41. After subtracting the total score of the reverse scored items from the total score of the flat items, the scale's own constant constant value of 50 is added to this score. The reliability (Kurder-Richardson Alpha) coefficient of the original version of the state anxiety scale was reported as 0.83-0.92, while the Turkish version was 0.94-0.96.

Stress ball Stress ball to be used; It is a 6 cm diameter, soft-textured, polyurethane ball, disinfected with a surface disinfectant.

Chewing gum The gum to be used is for all patients; the same brand is an easy-to-chew sugar-free gum that does not contain sorbitol and xylitol. Before the chewing gum was given to the patient, the hands of the patient and the researcher were disinfected with hand disinfectant. The gum was given to the patient in a package and he was allowed to open it himself.

Sphygmomanometer sphygmomanometer will be used for measurements. Pulse oximeter device Finger type pulse oximeter device will be used. The probe of the device, the hands of the patient and the researcher will be disinfected before and after each application.

Implementation of the Research and Collection of Data:

The consent of the individuals who met the inclusion criteria was obtained from the individuals who came to the blood collection outpatient clinic, and which group they would be included in will be determined by the researcher by drawing lots. First, the introductory data of the individual will be collected with the introduction form, and the arm diameter will be measured. Then, the initiative will be applied according to which group it will take place in.

Experiment 1 (stress ball) The patient will be asked to squeeze and loosen the stress ball with his non intervention hand for 5 minutes before and during the blood collection procedure. The researcher will continue to observe the patient to ensure that the stress ball is used throughout the blood collection procedure. After the blood collection procedure is completed, the patient will be referred to a nurse independent of the study to measure the patient's vital signs (blood pressure, pulse rate, SPO2 measurement and filling out the pain and anxiety scale). The nurse who made the last measurements will not know which group the patient is in. The nurse who made the final measurements will be blind.

Experiment 2 (Chewing gum) The patient will be given an unopened package of chewing gum and will be asked to chew the gum before and during the blood collection procedure.Chewing gum will take a total of 5 minutes. During this process, it will be observed by the researcher that the patient continues to chew gum.After the blood collection procedure is completed, the patient will be referred to a nurse independent of the study to measure the patient's vital signs (blood pressure, pulse rate, SPO2 measurement and filling out the pain and anxiety scale). The nurse who made the last measurements will not know which group the patient is in. The nurse who made the final measurements will be blind.

Control group Introductory form and introductory data will be obtained from the individuals they will be directed to the bloodletting nurse without any application. The same practices will be applied to the other two groups.

blood collection procedure

* Blood collection procedures will be done by a single nurse working in the blood collection unit. It will be ensured that the same nurse performs the intervention of all groups in order to avoid differences in the intervention due to the person performing the procedure.
* Blood collection will be done from the antecubital vein of the right or left arm in all patients.

After the application area is wiped with 70% alcohol and asepsis is achieved, blood will be drawn.

* Patients who will receive blood are individuals who come to donate blood at the request of a physician. Patients will not be subjected to any interventions such as taking extra blood, getting an examination, etc. for this research.
* In all applications, due to the Covid-19 process, attention will be paid to the use of masks and hand hygiene, ventilation of the environment and distance.

Distribution of the research Obtaining permissions for research; Hilal Türkben Polat, collection of data and the implementation of the initiative; Hilal Türkben Polat and Rukiye Burucu, introduction and method Rukiye Burucu, Hilal TÜRKBEN POLAT, findings and discussion Hilal Türkben Polat, Rukiye BURUCU.

Variables of the Study Dependent variables: Patient Post-procedure arterial blood pressure, heart rate, peripheral oxygen saturation, pain score, state anxiety score.

Independent variables: Patient: age, gender, body mass index (BMI), education level, marital status, employment status, income level, chronic disease status Ethical Dimension of Research Research permission was obtained from the XXX Ethics Committee (04.02.2022, 2022/3640), and application permission was obtained from XXX Hospital (25.11.2022 E-14567952-900-273749).

Limitations of the Research The limitation of the study is that the data of the study are collected from patients followed only in one center in Konya.

Evaluation of research data Statistics of the research will be done in SPSS 22 program; The data will be summarized as number, percentage, mean and standard deviation, chi-square analysis will be used to compare the sociodemographic characteristics of the experimental and control groups, and t-test for independent groups will be used for the means. The effect size obtained as a result of the calculations will be considered as ≤0.20 weak, if it is between 0.20<d<0.80, medium and d≥0.80 large effect size. The relationship between the scores will be examined by pearson correlation analysis, r≤0.25 is very weak in the evaluation of the correlation; 0.26≤ r ≤0.49 weak; 0.50≤ r ≤ 0.69 medium; 0.70≤ r ≤ 0.89 strong; If 0.90≤ r < 1, it will be considered very strong.

ELIGIBILITY:
Inclusion Criteria:

Being over 18 years old

* Having a body mass index of 30 and above
* Giving blood for analyzes upon the request of the physician
* Having the harmony of place and time
* Willingness to participate in the research

Exclusion Criteria:

* Absence of vision and hearing problems
* Presence of any disease that may affect pain perception
* Having cognitive problems
* Having a condition that prevents chewing gum
* Having a condition that prevents him from using the stress ball

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
pain severity | within 5 minutes after procedure
  The patient will be asked to evaluate the pain felt by the VAS pain scale.

SECONDARY OUTCOMES:
Anxiety state | within 5 minutes after procedure
  The level of anxiety felt by the patient will be evaluated with the anxiety scale.

OTHER OUTCOMES:
Arterial blood pressure value | within 5 minutes after procedure
  Measurement will be made with a manual sphygmomanometer;90/60 mmHg<blood pressure>140/90 mmHg
Heart rate value | "within 5 minutes after procedure
  It will be counted by resting from the apex with a stethoscope;60<heart rate>110
Oxygen saturation valu | within 5 minutes after procedure
  Measurement will be made with a pulse oximeter; saturation>95%

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan Univercity, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weijenberg RA, Lobbezoo F. Chew the Pain Away: Oral Habits to Cope with Pain and Stress and to Stimulate Cognition. Biomed Res Int. 2015;2015:149431. doi: 10.1155/2015/149431. Epub 2015 May 18. PMID 26090381
- [Result] Kabore RAF, Traore IA, Traore SIS, Bougouma CTHW, Augustin P, Ouro-Bang'na Maman AF. Broken needle during spinal anesthesia: an avoidable complication. Local Reg Anesth. 2018 Nov 23;11:111-113. doi: 10.2147/LRA.S175547. eCollection 2018. PMID 30538540
- [Result] Rodriguez-Calero MA, Blanco-Mavillard I, Morales-Asencio JM, Fernandez-Fernandez I, Castro-Sanchez E, de Pedro-Gomez JE. Defining risk factors associated with difficult peripheral venous Cannulation: A systematic review and meta-analysis. Heart Lung. 2020 May-Jun;49(3):273-286. doi: 10.1016/j.hrtlng.2020.01.009. Epub 2020 Feb 11. PMID 32057426
- [Result] Dat M, Jc TM, Ac N, Reis RK, Mh B, Sem T. Prevalence of and factors associated with difficult peripheral venipuncture in adult surgical patients. J Vasc Access. 2021 May;22(3):404-410. doi: 10.1177/1129729820939335. Epub 2020 Jul 28. PMID 32720556
- [Derived] Turkben Polat H, Burucu R. Effects of chewing gum and stress ball on pain and anxiety during blood collection in people with obesity: a randomized controlled study. Psychol Health Med. 2025 Nov 12:1-13. doi: 10.1080/13548506.2025.2587975. Online ahead of print. PMID 41222481